CLINICAL TRIAL: NCT00654862
Title: Randomized Controlled, Double-Blind, Sample Size-Calculated, Three-Period Crossover, Phase 1 Study to Investigate the Efficacy of a Single Oral Dose of Cocoa Phenols on Blood, Pressure, Heart Rate and Plasma Levels of Phenols, Bioactive Nitric Oxide and Oxidation Markers in Subjects With Stage 1 Essential Hypertension and Optimal Blood Pressure
Brief Title: Acute Hemodynamic Effects of Cocoa Polyphenols in Subjects With Hypertension and Optimal Blood Pressure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Dirk Taubert, University of Cologne
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ECA-02-006
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Subjects with stage 1 hypertension
  Interventions: Dietary Supplement: cocoa polyphenols
- 2 (Experimental): Subjects with optimal blood pressure
  Interventions: Dietary Supplement: cocoa polyphenols

INTERVENTIONS:
Dietary Supplement: cocoa polyphenols — Oral administration of capsules with 1000 mg polyphenols, 250 mg polyphenols or placebo
  Arms: 1
Dietary Supplement: cocoa polyphenols — Oral administration of capsules with 1000 mg polyphenols, 250 mg polyphenols or placebo
  Arms: 2

SUMMARY:
Intake of cocoa-containing foods has been found to lower blood pressure (BP) in several clinical trials. It is supposed that the cocoa polyphenols represent the active principle, lowering BP by increasing the formation of vasodilative nitric oxide. However, direct evidence for this assumption from controlled clinical studies is lacking. Moreover, in hypertensive subjects vascular dilation appears to be impaired due to endothelial dysfunction and vascular smooth muscle remodeling, but it is unclear whether the BP response to cocoa phenols differs between subjects with high blood pressure and optimal blood pressure.

The investigators hypothesized that (1) intake of cocoa phenols cause a dose-dependent, acute elevation of circulating bioactive NO levels and a reduction in BP, and that (2) the NO elevation and BP reduction are impaired in patients with hypertension.

To test this hypothesis, the investigators will conduct a prospective, randomized, placebo-controlled, double-blind, sample size-calculated, three-period crossover study with pre-planned statistical analysis and trial monitoring, in which cocoa phenols will be orally administered to subjects with mild essential hypertension or subjects with optimal blood pressure. The effects on blood pressure, heart rate, arterial function and plasma levels of cocoa phenols, circulating bioactive nitric oxide, and plasma markers of oxidative stress will be evaluated. After a 7-day cocoa-free run-in period and a 12-hour overnight fast, 48 subjects (24 with hypertension and 24 sex-, and age (+/- 2yrs)-matched subjects with optimal blood pressure) will receive either a single dose of 1000 mg cocoa polyphenols, 250 mg cocoa phenols or placebo (in capsules of equal form and weight). Each intervention will be followed by a 7-day cocoa-free washout period before cross-over to the subsequent intervention. Subjects will be allocated to the intervention sequence by permuted block randomization (i.e. permuted blocks of 2 subjects with high BP and 2 subjects with optimal BP each, are assigned to permutations of the tree interventions). Measurements of hemodynamic and plasma parameters will be performed directly before and 30, 60, 90, 120, 180, 300, and 480 min after capsule administration. Included subjects will be counseled to maintain their usual diet and physical activity and to abstain from all cocoa products during the study. Analysis of the data will be performed on an intention-to-treat basis.

ELIGIBILITY:
Inclusion Criteria:

* Unpaid volunteers of both sex between 50 and 75 years of age in good general health.
* Diagnosis of stage 1 essential hypertension (BP between 140/90 and 160/100 mmHg) or optimal BP below 120/80) and stable BP values.
* No antihypertensive medications or nutritional supplements.
* Non-manual workers or pensioners of higher socioeconomic status (household income of more than 20,000 €/year)
* Leisure physical activity of less than 7 METs per week
* Normal levels of plasma lipids and plasma glucose.

Exclusion Criteria:

* Cardiovascular diseases (other than hypertension).
* Diabetes mellitus.
* Hyper-/dyslipidemia.
* Gastrointestinal diseases
* Hepatic and renal disorders
* Pulmonary diseases.
* Coagulopathy.
* Cancer.
* Psychiatric disorders.
* Alcohol or drug dependence.
* Seizure disorders.
* History of organ transplantation.
* Surgery within the last 12 months.
* Positive tests for HIV, hepatitis B or C.
* Body-mass index of more than 27.5 or less than 18.5 kg/m2
* Active smokers of tobacco within the last five years.
* Regular users of medications.
* Use of any medication within the last two weeks before entry.
* Users of vitamin, mineral or polyphenol supplements or other bioactive food supplements.
* Regular consumers of chocolate or other cocoa products of more than 1 serving per week.
* Subjects will be excluded if they are unable to give informed consent for all procedures. Subjects who are not capable or willing to attend to all interventions will be withdrawn.
* Subjects will be withdrawn if the allocation concealment is disclosed.
* Subjects will be withdrawn if any adverse events requiring further monitoring or medical treatment occur.
* A systolic BP >170 mmHg or <100 mmHg or a diastolic BP >110 mmHg or <50 mmHg at a single determination will result in immediate withdrawal of the participant from the study and the appropriate treatment will be resumed.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-10; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Change in systolic and diastolic blood pressure | Assessments at 3 time points

SECONDARY OUTCOMES:
Changes in plasma levels of bioactive nitric oxide, arterial function, oxidation markers and cocoa polyphenols | Assessments at 3 time points

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Taubert, MD, PhD, Principal Investigator — University of Cologne
Locations (1):
- Department of Pharmacology, University of Cologne, Cologne, Germany

REFERENCES:
- [Background] Taubert D, Roesen R, Lehmann C, Jung N, Schomig E. Effects of low habitual cocoa intake on blood pressure and bioactive nitric oxide: a randomized controlled trial. JAMA. 2007 Jul 4;298(1):49-60. doi: 10.1001/jama.298.1.49. PMID 17609490
- [Background] Taubert D, Berkels R, Roesen R, Klaus W. Chocolate and blood pressure in elderly individuals with isolated systolic hypertension. JAMA. 2003 Aug 27;290(8):1029-30. doi: 10.1001/jama.290.8.1029. No abstract available. PMID 12941673